CLINICAL TRIAL: NCT04154189
Title: A Multicenter, Open-label, Randomized Phase 2 Study to Compare the Efficacy and Safety of Lenvatinib in Combination With Ifosfamide and Etoposide Versus Ifosfamide and Etoposide in Children, Adolescents and Young Adults With Relapsed or Refractory Osteosarcoma (OLIE)
Brief Title: A Study to Compare the Efficacy and Safety of Ifosfamide and Etoposide With or Without Lenvatinib in Children, Adolescents and Young Adults With Relapsed and Refractory Osteosarcoma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Eisai Inc. (Industry)
Collaborators: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: E7080-G000-230; 2019-003696-19 (EudraCT Number)
Record Dates: First submitted 2019-11-01; First posted 2019-11-06 (Actual); Results first posted 2023-08-07 (Actual); Last update posted 2024-07-22 (Actual); Status verified 2024-07

CONDITIONS: Osteosarcoma
Keywords: Osteosarcoma; Lenvatinib; Ifosfamide; Etoposide; E7080; Relapsed or Refractory Osteosarcoma; Pediatrics; Chemotherapy
MeSH Terms: conditions — Osteosarcoma; Recurrence | interventions — lenvatinib; Ifosfamide; Etoposide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Randomization Phase: Lenvatinib + Ifosfamide + Etoposide (Experimental): Participants with relapsed or refractory osteosarcoma will receive lenvatinib in combination with ifosfamide and etoposide.
  Interventions: Drug: Lenvatinib; Drug: Ifosfamide; Drug: Etoposide
- Randomization Phase: Ifosfamide + Etoposide (Active Comparator): Participants with relapsed or refractory osteosarcoma will receive ifosfamide with etoposide. Participants with relapsed or refractory osteosarcoma may receive optional lenvatinib plus or minus chemotherapy (Ifosfamide and Etoposide) if disease progression is observed in study.
  Interventions: Drug: Ifosfamide; Drug: Etoposide; Drug: Lenvatinib

INTERVENTIONS:
Drug: Lenvatinib — Lenvatinib 14 milligrams per square meter (mg/m^2) capsules will be administered once daily on Days 1 to 21 of each 21-day cycle until disease progression (PD), development of unacceptable toxicity, participant request, withdrawal of consent, or discontinuation of study by the sponsor.
  An extemporaneous suspension of lenvatinib capsules may be used for participants unable to swallow capsules.
  Other Names: E7080
  Arms: Randomization Phase: Lenvatinib + Ifosfamide + Etoposide
Drug: Ifosfamide — Ifosfamide 3000 milligrams per square meter per day (mg/m^2/day) intravenous infusion will be administered on Days 1 to 3 of each 21-day cycle for a total of 5 cycles.
Drug: Etoposide — Etoposide 100 mg/m^2/day intravenous infusion will be administered on Days 1 to 3 of each 21-day cycle for a total of 5 cycles.
Drug: Lenvatinib — Lenvatinib 14 mg/m^2 capsules will be administered once daily on Days 1 to 21 of each 21-day cycle until the next PD (per response evaluation criteria in solid tumors [RECIST] 1.1 as assessed by investigator), development of unacceptable toxicity, participant request, or withdrawal of consent, whichever occurs first.
  Other Names: E7080
  Arms: Randomization Phase: Ifosfamide + Etoposide

SUMMARY:
This Is a Multicenter, Randomized, Open-Label, Parallel-Group, Phase 2 Study to Compare the Efficacy and Safety of Lenvatinib in Combination with Ifosfamide and Etoposide Versus Ifosfamide and Etoposide in Children, Adolescents, and Young Adults with Relapsed or Refractory Osteosarcoma.

ELIGIBILITY:
Inclusion Criteria:

1. Histologically or cytologically confirmed diagnosis of high grade osteosarcoma
2. Refractory or relapsed osteosarcoma after 1 to 2 prior lines of systemic treatments
3. Measurable or evaluable disease per RECIST 1.1.
4. Life expectancy of 12 weeks or more
5. Lansky play score greater than or equal to (>=) 50 Percent (%) or Karnofsky Performance Status score >=50%. Use Karnofsky for participants >=16 years of age and Lansky for participants less than (<)16 years of age. Participants who are unable to walk because of paralysis, but who are able to perform activities of daily living while wheelchair bound, will be considered ambulatory for the purpose of assessing the performance score
6. Adequate organ function per blood work
7. Adequate cardiac function as evidenced by left ventricular ejection fraction (LVEF) >=50% at baseline as determined by echocardiography or multigated acquisition (MUGA) scan
8. Adequately controlled blood pressure (BP) with or without antihypertensive medications, defined as:

   BP <95th percentile for sex, age, and height/length at screening (as per National Heart Lung and Blood Institute guidelines) and no change in antihypertensive medications within 1 week prior to Cycle 1 Day 1. Participants >18 years of age should have BP less than or equal to (<=) 150/90 millimeters of Mercury at screening and no change in antihypertensive therapy within 1 week prior to Cycle 1 Day 1
9. Washout before Cycle 1 Day 1 of 3 weeks in case of prior chemotherapy, 6 weeks if treatment included nitrosoureas; 4 weeks for definitive radiotherapy, 2 weeks for palliative radiotherapy; and 3 months from high-dose chemotherapy and stem cell rescue. For all other anti-cancer therapies, washout before Cycle 1 Day 1 of at least 5 half-lives (or at least 28 days, whichever is shorter). Participants must have recovered [to Grade <=1, except for alopecia, ototoxicity, and Grade <=2 peripheral neuropathy, per common terminology criteria for adverse events (CTCAE) v5.0] from the acute toxic effects of all prior anticancer therapy before Cycle 1 Day 1
10. Must have no prior history of lenvatinib treatment

Eligibility for optional lenvatinib crossover:

1. Disease progression per RECIST 1.1 (as confirmed by IIR for all participants who crossover prior to the study data-cut)
2. No new systemic anti-cancer medication administered after the last dose of study drugs
3. Meets all safety parameters listed in the inclusion criteria and none listed in the exclusion criteria
4. Study is ongoing

Exclusion Criteria:

1. Any active infection or infectious illness unless fully recovered prior to Cycle 1 Day 1 (that is, no longer requiring systemic treatment)
2. Participants with central nervous system metastases are not eligible, unless they have completed local therapy (example, whole brain radiation therapy, surgery or radiosurgery) and have discontinued the use of corticosteroids for this indication for at least 2 weeks before Cycle 1 Day 1
3. Active second malignancy within 2 years prior to enrollment ([in addition to osteosarcoma], but not including definitively treated superficial melanoma, carcinoma-in-situ, basal or squamous cell carcinoma of the skin)
4. Has had major surgery within 3 weeks prior to Cycle 1 Day 1. Note: Adequate wound healing after major surgery must be assessed clinically, independent of time elapsed for eligibility
5. A clinically significant electrocardiogram (ECG) abnormality, including a marked baseline prolonged QT or corrected QT (QTc) interval (example, a repeated demonstration of a QTc interval greater than [>] 480 millisecond [msec])
6. Has clinically significant cardiovascular disease within 6 months from first dose of study intervention, including New York Heart Association Class III or IV congestive heart failure, unstable angina, myocardial infarction, cerebral vascular accident, or cardiac arrhythmia associated with hemodynamic instability. Note: Medically controlled arrhythmia would be permitted
7. Gastrointestinal malabsorption, gastrointestinal anastomosis, or any other condition that in the opinion of the investigator might affect the absorption of lenvatinib
8. Pre-existing Grade >=3 gastrointestinal or non-gastrointestinal fistula
9. Gastrointestinal bleeding or active hemoptysis (bright red blood of at least 1 divided [/] by 2 teaspoon) within 3 weeks prior to Cycle 1 Day 1
10. Radiographic evidence of intratumoral cavitation, encasement, or invasion of a major blood vessel. Additionally, the degree of proximity to major blood vessels should be considered for exclusion because of the potential risk of severe hemorrhage associated with tumor shrinkage/necrosis after lenvatinib therapy
11. History of ifosfamide-related Grade >=3 nephrotoxicity or encephalopathy
12. Known to be human immunodeficiency virus (HIV) positive
13. Known active Hepatitis B (example, Hepatitis B surface antigen [HBsAg] reactive) or Hepatitis C (example, hepatitis C virus [HCV] ribonucleic acid [RNA] [qualitative] is detected). Note: Testing for Hepatitis B or Hepatitis C is required at screening only when mandated by local health authority

Ages: 2 Years to 25 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 81 (Actual)
Dates: Start 2020-03-23 (Actual); Primary Completion 2022-06-22 (Actual); Study Completion 2023-08-17 (Actual)

CONTACTS AND LOCATIONS:
Locations (84):
- United States (16):
  - Children's of Alabama, Birmingham, Alabama
  - Loma Linda University Medical Center, Loma Linda, California
  - Children's Hospital of Orange County, Orange, California
  - UCSF Benioff Children's Hospitals, San Francisco, California
  - Childrens Hospital Colorado, Aurora, Colorado
  - Children's National Medical Center, Washington D.C., District of Columbia
  - Riley Hospital For Children, Indianapolis, Indiana
  - Dana Farber Cancer Institute, Boston, Massachusetts
  - University of Mississippi Medical Center, Jackson, Mississippi
  - Hackensack University Medical Center, Hackensack, New Jersey
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - Cincinnati Children's Hospital Medical Center, Cincinnati, Ohio
  - Vanderbilt University Medical Center, Nashville, Tennessee
  - Children's Medical Center Dallas, Dallas, Texas
  - Cook Children's Health Care System, Fort Worth, Texas
  - Texas Children's Hospital, Houston, Texas
- Australia (5):
  - Chris O'Brien Lifehouse Hospital, Camperdown
  - Perth Childrens Hospital, Nedlands
  - Royal Children's Hospital Melbourne, Parkville
  - Queensland Children's Hospital, South Brisbane
  - Children's Hospital at Westmead, Westmead
- St. Anna Kinderspital, Vienna, Austria
- UZ Gent, Ghent, Belgium
- Hospital For Sick Children, Toronto, Canada
- Czechia (2):
  - FN Brno 2 Detska Klinika, Brno
  - Fakultní nemocnice v Motole, Prague
- Tampereen yliopistollinen sairaala, Tampere, Länsi-Suomen Lääni, Finland
- France (12):
  - Centre Hospitalier Universitaire de Bordeaux, Hopital Pellegrin, Bordeaux
  - Centre Oscar Lambret, Lille
  - Centre Léon Berard, Lyon
  - Hopitaux de La Timone, Marseille
  - Hôpital de La Mère Et de L'enfant, Nantes
  - CHU de Nice, Nice
  - Hôpital Armand Trousseau, Paris
  - Institut Curie, Paris
  - Hopital de Hautepierre, Strasbourg
  - Hôpital Des Enfants, Toulouse
  - CHRU Nancy, Vandœuvre-lès-Nancy
  - Institut Gustave Roussy, Villejuif
- Hong Kong (2):
  - Hong Kong Children's Hospital, Hong Kong
  - Prince of Wales Hospital, Hong Kong
- Children's Health Ireland at Crumlin, Dublin, Ireland
- Schneider Children's Medical Center of Israel, Petah Tikva, Israel
- Italy (5):
  - Istituti Ortopedici Rizzoli, Bologna
  - Azienda Ospedaliera A Meyer, Florence
  - Istituto Giannina Gaslini, Genova
  - Istituto Nazionale Dei Tumori, Milan
  - IRCCS Ospedale Pediatrico Bambino Gesù, Roma
- Princess Maxima Center for Pediatric Oncology, Utrecht, Netherlands
- New Zealand (2):
  - Auckland City Hospital, Auckland
  - Starship Children's Hospital, Auckland
- Singapore (3):
  - KK Women's and Children's Hospital, Singapore
  - National Cancer Centre, Singapore
  - National University Hospital, Singapore
- South Korea (5):
  - National Cancer Center, Goyang-si
  - Asan Medical Center, Seoul
  - Samsung Medical Center, Seoul
  - Seoul National University Hospital, Seoul
  - Severance Hospital Yonsei University Health System, Seoul
- Spain (8):
  - Hospital Universitario de Cruces, Barakaldo
  - Hospital Sant Joan de Deu, Barcelona
  - Hospital Universitario Vall d'Hebrón, Barcelona
  - Hospital Infantil Universitario Niño Jesus, Madrid
  - Hospital Universitario Fundacion Jimenez Diaz, Madrid
  - Hospital Universitario La Paz, Madrid
  - Hospital Universitario Virgen del Rocio, Seville
  - Hospital Universitari i Politecnic La Fe de Valencia, Valencia
- Sweden (3):
  - Drottning Silvias Barn Och Ungdomssjukhus, Gothenburg
  - Skanes Universitetssjukhus Lund, Lund
  - Karolinska Universitetssjukhuset Solna, Stockholm
- Switzerland (2):
  - Centre Hospitalier Universitaire Vaudois, Lausanne
  - Kinderspital Zürich - Eleonorenstiftung, Zurich
- Taiwan (2):
  - National Taiwan University Hospital, Taipei
  - Taipei Veterans General Hospital, Taipei
- United Kingdom (10):
  - Birmingham Children's Hospital, Birmingham
  - The Royal Hospital for Children, Bristol
  - Royal Hospital for Children, Glasgow
  - Leeds Children Hospital, Leeds
  - Alder Hey Children's Hospital, Liverpool
  - UCL Cancer Institute, London
  - Royal Manchester Childrens Hospital, Manchester
  - The Christie NHS Foundation Trust, Manchester
  - Royal Victoria Infirmary, Newcastle
  - John Radcliffe Hospital, Oxford

IPD SHARING:
Plan to Share IPD: Yes
Eisai's data sharing commitment and further information on how to request data can be found on our website http://eisaiclinicaltrials.com/.

REFERENCES:
- [Derived] Gaspar N, Hung GY, Strauss SJ, Campbell-Hewson Q, Dela Cruz FS, Glade Bender JL, Koh KN, Whittle SB, Chan GC, Gerber NU, Palmu S, Morgenstern DA, Longhi A, Baecklund F, Lee JA, Locatelli F, Marquez Vega C, Janeway KA, McCowage G, McCabe MG, Bidadi B, Huang J, McKenzie J, Okpara CE, Bautista F; OLIE Study Investigators. Lenvatinib Plus Ifosfamide and Etoposide in Children and Young Adults With Relapsed Osteosarcoma: A Phase 2 Randomized Clinical Trial. JAMA Oncol. 2024 Dec 1;10(12):1645-1653. doi: 10.1001/jamaoncol.2024.4381. PMID 39418029
- [Derived] Gaspar N, Venkatramani R, Hecker-Nolting S, Melcon SG, Locatelli F, Bautista F, Longhi A, Lervat C, Entz-Werle N, Casanova M, Aerts I, Strauss SJ, Thebaud E, Morland B, Nieto AC, Marec-Berard P, Gambart M, Rossig C, Okpara CE, He C, Dutta L, Campbell-Hewson Q. Lenvatinib with etoposide plus ifosfamide in patients with refractory or relapsed osteosarcoma (ITCC-050): a multicentre, open-label, multicohort, phase 1/2 study. Lancet Oncol. 2021 Sep;22(9):1312-1321. doi: 10.1016/S1470-2045(21)00387-9. Epub 2021 Aug 17. PMID 34416158
- [Derived] Gaspar N, Campbell-Hewson Q, Huang J, Okpara CE, Bautista F. OLIE, ITCC-082: a Phase II trial of lenvatinib plus ifosfamide and etoposide in relapsed/refractory osteosarcoma. Future Oncol. 2021 Nov;17(32):4249-4261. doi: 10.2217/fon-2021-0743. Epub 2021 Aug 12. PMID 34382412

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants took part in the study at 84 investigative sites in Austria, Australia, Belgium, Hong Kong, Korea, New Zealand, Singapore, Taiwan, Czech Republic, Finland, France, Israel, Ireland, Italy, Netherlands, Spain, Sweden, Switzerland, United Kingdom, Canada, and the United States.
Pre-assignment Details: A total of 99 participants were screened, 18 failed screening. 81 participants were enrolled and randomized, out of which 78 received the study treatment.
Groups:
- Treatment Arm A: Lenvatinib + Ifosfamide + Etoposide: Participants received lenvatinib 14 milligrams per square meter (mg/m^2), capsules, orally, once daily, plus ifosfamide 3000 milligrams per square meter per day (mg/m^2/day), intravenously and etoposide 100 mg/m^2/day, intravenously. Ifosfamide and etoposide were administered on Days 1 to 3 of each 21-day cycle for up to 5 cycles. Lenvatinib was administered in continuous 21-day cycles. Treatment continued until disease progression (PD), development of unacceptable toxicity, participant choice, withdrawal of consent or discontinuation of study by the sponsor, whichever occurred first.
- Treatment Arm B: Ifosfamide + Etoposide: Participants received ifosfamide 3000 mg/m^2/day, intravenously and etoposide 100 mg/m^2/day, intravenously on Days 1 to 3 of each 21-day cycle for up to 5 cycles. Participants who had PD per response evaluation criteria in solid tumors (RECIST) version (v) 1.1 were eligible for an optional lenvatinib treatment (14 mg/m^2, capsules, orally, once daily in continuous 21-day cycles until next PD, development of unacceptable toxicity, participant choice, withdrawal of consent or discontinuation of study by the sponsor, whichever occurred first) plus any remaining cycles of chemotherapy if 5 cycles were not completed prior to PD.
Period: Overall Study
Arm/Group | Treatment Arm A: Lenvatinib + Ifosfamide + Etoposide | Treatment Arm B: Ifosfamide + Etoposide
Started (Participant Flow (including deaths in reasons of discontinuation) was based on Full Analysis Set (Full Analysis Set included all randomized participants regardless of the treatment actually received).) | 40 | 41
Treated (Safety Analysis Set) | 39 | 39
Optional Lenvatinib Treatment (Arm B Only) (Participants from Treatment Arm B: Ifosfamide + Etoposide who had PD per RECIST v1.1 were eligible to receive an optional lenvatinib treatment plus any remaining cycles of chemotherapy (ifosfamide + etoposide) if 5 cycles were not completed prior to PD.) | 0 | 16
Completed | 0 | 0
Not Completed | 40 | 41
Not completed — Withdrawal by Subject | 4 | 6
Not completed — Survival follow-up discontinued by sponsor | 8 | 10
Not completed — Participants transitioned to patient access program (PAP) | 1 | 0
Not completed — Participants transitioned to managed access program (MAP) | 2 | 0
Not completed — Death | 25 | 25

BASELINE CHARACTERISTICS:
Population: Full Analysis Set (FAS) included all randomized participants regardless of the treatment actually received.
Groups:
- Treatment Arm A: Lenvatinib + Ifosfamide + Etoposide: Participants received lenvatinib 14 mg/m^2, capsules, orally, once daily, plus ifosfamide 3000 mg/m^2/day, intravenously and etoposide 100 mg/m^2/day, intravenously. Ifosfamide and etoposide were administered on Days 1 to 3 of each 21-day cycle for up to 5 cycles. Lenvatinib was administered in continuous 21-day cycles. Treatment continued until PD, development of unacceptable toxicity, participant choice, withdrawal of consent or discontinuation of study by the sponsor, whichever occurred first.
- Treatment Arm B: Ifosfamide + Etoposide: Participants received ifosfamide 3000 mg/m^2/day, intravenously and etoposide 100 mg/m^2/day, intravenously on Days 1 to 3 of each 21-day cycle for up to 5 cycles. Participants who had PD per RECIST v1.1 were eligible for an optional lenvatinib treatment (14 mg/m^2, capsules, orally, once daily in continuous 21-day cycles until next PD, development of unacceptable toxicity, participant choice, withdrawal of consent or discontinuation of study by the sponsor, whichever occurred first) plus any remaining cycles of chemotherapy if 5 cycles were not completed prior to PD.
- Total: Total of all reporting groups
Arm/Group | Treatment Arm A: Lenvatinib + Ifosfamide + Etoposide | Treatment Arm B: Ifosfamide + Etoposide | Total
Number analyzed (Participants) | 40 | 41 | 81
Age, Continuous [Mean (Standard Deviation); unit: years] | 15.6 (3.76) | 14.3 (4.16) | 14.9 (3.99)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 15 | 20 | 35
  Male | 25 | 21 | 46
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2 | 3 | 5
  Not Hispanic or Latino | 38 | 33 | 71
  Unknown or Not Reported | 0 | 5 | 5
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 24 | 26 | 50
  Black or African American | 1 | 1 | 2
  Asian | 13 | 7 | 20
  American Indian or Alaskan Native | 0 | 1 | 1
  Other | 2 | 4 | 6
  Missing | 0 | 2 | 2

OUTCOME MEASURES:

1. Primary Outcome: Progression-free Survival (PFS) by Independent Imaging Review (IIR) Assessment
Description: PFS as assessed by IIR was defined as the time from the date of randomization to the date of the first documentation of PD or date of death (whichever occurred first), as determined using RECIST v1.1. PD was defined as at least a 20 percent (%) increase or 5 millimeter (mm) increase in the sum of diameters of target lesions (taking as reference the smallest sum on study) recorded since the treatment started or the appearance of 1 or more new lesions. PFS was analyzed using Kaplan-Meier method.
Time Frame: From the date of randomization to the date of the first documentation of PD or date of death, whichever occurred first (up to 20.5 months)
Population: FAS included all randomized participants regardless of the treatment actually received.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Treatment Arm A: Lenvatinib + Ifosfamide + Etoposide | Treatment Arm B: Ifosfamide + Etoposide
Number analyzed (Participants) | 40 | 41
months | 6.5 [5.7 to 8.2] | 5.5 [2.9 to 6.5]
Statistical Analysis 1: Comparison: Treatment Arm A: Lenvatinib + Ifosfamide + Etoposide vs Treatment Arm B: Ifosfamide + Etoposide; Test type: Superiority; p = 0.0396, Log Rank — One-sided P value; Hazard Ratio (HR) = 0.54, 95% CI 2-sided [0.27 to 1.08] — Hazard ratio was based on Cox Proportional Hazard Model including treatment group as a factor and stratified by Age (less than [<]18 years, more than or equal to [>=]18 years) in interactive response technology (IRT). Efron method was used for ties

2. Secondary Outcome: Percentage of Participants With PFS at Month 4 (PFS-4m Rate) by IIR Assessment
Description: PFS rate at 4 months as assessed by IIR was defined as the percentage of participants who were alive and without PD at 4 months from the randomization date using RECIST v1.1. PD was defined as at least a 20% increase or 5 mm increase in the sum of diameters of target lesions (taking as reference the smallest sum on study) recorded since the treatment started or the appearance of 1 or more new lesions. The PFS-4m was estimated using the Kaplan-Meier method.
Time Frame: Month 4
Population: FAS included all randomized participants regardless of the treatment actually received.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Treatment Arm A: Lenvatinib + Ifosfamide + Etoposide | Treatment Arm B: Ifosfamide + Etoposide
Number analyzed (Participants) | 40 | 41
percentage of participants | 76.3 [59.3 to 86.9] | 66.0 [47.7 to 79.2]
Statistical Analysis 1: Comparison: Treatment Arm A: Lenvatinib + Ifosfamide + Etoposide vs Treatment Arm B: Ifosfamide + Etoposide; Test type: Other — Difference in PFS rates, and 2-sided 95% confidence intervals (CIs): CI and p-value constructed using the difference of the 2 Kaplan-Meier PFS rates (4 months) and the 2 corresponding Greenwood standard errors; p = 0.1683, Kaplan-Meier Method — One-sided P value; Difference in Percentage = 10.2, 95% CI 2-sided [-10.6 to 31.1]

3. Secondary Outcome: Percentage of Participants With PFS at 1 Year or Month 12 (PFS-1y Rate) by IIR Assessment
Description: PFS-1y rate as assessed by IIR was defined as the percentage of participants who were alive and without PD at 1 year from randomization date using RECIST v1.1. PD was defined as at least a 20% increase or 5 mm increase in the sum of diameters of target lesions (taking as reference the smallest sum on study) recorded since the treatment started or the appearance of 1 or more new lesions. PFS-1y rate was estimated using Kaplan-Meier method.
Time Frame: Month 12 or 1 Year
Population: FAS included all randomized participants regardless of the treatment actually received.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Treatment Arm A: Lenvatinib + Ifosfamide + Etoposide | Treatment Arm B: Ifosfamide + Etoposide
Number analyzed (Participants) | 40 | 41
percentage of participants | NA [NA to NA] — Number and 95% confidence interval data could not be estimated because all participants had an event or were censored before Month 12. | 14.9 [1.1 to 44.5]

4. Secondary Outcome: Overall Survival (OS)
Description: OS was defined as the time from the date of randomization to the date of death from any cause. The median OS was from Kaplan-Meier product-limit estimates and 2-sided 95% CIs from a generalized Brookmeyer and Crowley method.
Time Frame: From the date of randomization to the date of death from any cause (up to 37.1 months)
Population: FAS included all randomized participants regardless of the treatment actually received.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Treatment Arm A: Lenvatinib + Ifosfamide + Etoposide | Treatment Arm B: Ifosfamide + Etoposide
Number analyzed (Participants) | 40 | 41
months | 12.4 [10.4 to 19.8] | 17.2 [11.1 to 22.3]
Statistical Analysis 1: Comparison: Treatment Arm A: Lenvatinib + Ifosfamide + Etoposide vs Treatment Arm B: Ifosfamide + Etoposide; Test type: Other; p = 0.3924, Stratified Log-rank One-sided Test — Nominal p-value from stratified log-rank test adjusted for the randomization stratification factor, that is, age; Hazard Ratio (HR) = 0.93, 95% CI 2-sided [0.53 to 1.62] — Hazard ratio was based on a Cox Proportional Hazard Model including treatment group as a factor and stratified by Age (<18 years, >=18 years) in IRT. Efron method was used for ties

5. Secondary Outcome: Percentage of Participants With Overall Survival at 1 Year or Month 12 (OS-1y)
Description: OS-1y was defined as the time from the date of randomization to the date of death from any cause assessed up to 1 year. OS was calculated using the Kaplan-Meier method.
Time Frame: Month 12 or 1 Year
Population: FAS included all randomized participants regardless of the treatment actually received.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Treatment Arm A: Lenvatinib + Ifosfamide + Etoposide | Treatment Arm B: Ifosfamide + Etoposide
Number analyzed (Participants) | 40 | 41
percentage of participants | 49.2 [28.5 to 67.0] | 72.1 [54.2 to 83.9]
Statistical Analysis 1: Comparison: Treatment Arm A: Lenvatinib + Ifosfamide + Etoposide vs Treatment Arm B: Ifosfamide + Etoposide; Test type: Other — Difference and 95% CI: difference of 2 Kaplan-Meier OS-1y rates and corresponding Greenwood standard errors; p = 0.0352, Kaplan Meier Method — One-sided P value; Difference in Percentage = -22.9, 95% CI 2-sided [-47.6 to 1.9]

6. Secondary Outcome: Objective Response Rate at Month 4 (ORR-4m) by IIR Assessment
Description: ORR-4m was defined as the percentage of participants with best overall response of complete response (CR) or partial response (PR) as determined by IIR using RECIST v1.1 within the first 4 months. CR: defined as the disappearance of all target and non-target lesions (non-lymph nodes). All pathological lymph nodes (whether target or non-target) must have a reduction in their short axis to less than (<) 10 mm. PR: defined as at least a 30% decrease in the sum of diameters of target lesions, taking as reference the baseline sum diameters. 95% confidence interval (CI) of ORR was calculated using the method of Clopper and Pearson.
Time Frame: Month 4
Population: FAS included all randomized participants regardless of the treatment actually received.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Treatment Arm A: Lenvatinib + Ifosfamide + Etoposide | Treatment Arm B: Ifosfamide + Etoposide
Number analyzed (Participants) | 40 | 41
percentage of participants | 15.0 [5.7 to 29.8] | 7.3 [1.5 to 19.9]
Statistical Analysis 1: Comparison: Treatment Arm A: Lenvatinib + Ifosfamide + Etoposide vs Treatment Arm B: Ifosfamide + Etoposide; Test type: Other — Difference calculated as Treatment Arm A: Lenvatinib + Ifosfamide + Etoposide minus Treatment Arm B: Ifosfamide + Etoposide. 2-sided 95% CI: Miettinen-Nurminen (Score) confidence limits, stratified by randomization stratification factor age (<18 and >=18 years); Difference in Percentage = 7.7, 95% CI 2-sided [-6.4 to 22.3]

7. Secondary Outcome: ORR by IIR Assessment
Description: ORR by IIR was defined as the percentage of participants with best overall response of CR or PR determined using RECIST v1.1. CR: defined as the disappearance of all target and non-target lesions (non-lymph nodes). All pathological lymph nodes (whether target or non-target) must have a reduction in their short axis to <10 mm. PR: defined as at least a 30% decrease in the sum of diameters of target lesions, taking as reference the baseline sum diameters. 95% CI of ORR was calculated using the method of Clopper and Pearson.
Time Frame: From the date of randomization to the date of the first documentation of CR or PR (up to 20.5 months)
Population: FAS included all randomized participants regardless of the treatment actually received.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Treatment Arm A: Lenvatinib + Ifosfamide + Etoposide | Treatment Arm B: Ifosfamide + Etoposide
Number analyzed (Participants) | 40 | 41
percentage of participants | 15.0 [5.7 to 29.8] | 9.8 [2.7 to 23.1]
Statistical Analysis 1: Comparison: Treatment Arm A: Lenvatinib + Ifosfamide + Etoposide vs Treatment Arm B: Ifosfamide + Etoposide; Test type: Other — [test comment as in outcome 6, analysis 1]; Difference in Percentage = 5.2, 95% CI 2-sided [-10.3 to 20.0]

8. Secondary Outcome: Number of Participants With Treatment-emergent Adverse Events (TEAEs) and Treatment-emergent Serious Adverse Events (TESAEs)
Description: TEAE was defined as an adverse event (AE) that emerged during time from first dose to 30 days following last dose of drug, having been absent at pretreatment or reemerged during treatment, having been present at pretreatment but stopped before treatment, or worsened in severity during treatment relative to pretreatment state, when AE was continuous. Serious adverse events (SAE) was defined as untoward medical occurrence that at any dose resulted in death; was life threatening; resulted in persistent or significant disability; was congenital anomaly or medically important due to other reasons than above mentioned criteria.
Time Frame: From first dose up to 30 days after the last dose of study drug (up to 40.8 months)
Population: Safety Analysis Set included participants who received at least 1 dose of any study drug.
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment Arm A: Lenvatinib + Ifosfamide + Etoposide | Treatment Arm B: Ifosfamide + Etoposide
Number analyzed (Participants) | 39 | 39
Participants
  Participants with TEAEs | 38 | 39
  Participants with TESAEs | 30 | 20

9. Secondary Outcome: Treatment Arm A: Plasma Concentration of Lenvatinib
Description: Plasma concentration of lenvatinib in participants from Treatment Arm A (Lenvatinib + Ifosfamide + Etoposide) at different time points were reported. As planned, data for this outcome measure was analyzed for treatment arm A only. Lenvatinib concentration in plasma was quantified using a validated liquid chromatography tandem mass spectrometry (LC-MS/MS) method.
Time Frame: Cycle 1 Day 1: 0.5-4 hours and 6-10 hours post-dose; Cycle 1 Day 15: Pre-dose, 0.5-4 hours and 6-10 hours post-dose; Cycle 2 Day 1: Pre-dose (each Cycle length = 21 days)
Population: Population Pharmacokinetic (PK) Analysis Set included those participants who received at least 1 dose of lenvatinib and had documented dose administration history and measurable plasma concentrations of lenvatinib. Here "overall number of participants analyzed, N" signifies participants who were evaluable for this outcome measure. Here "number analyzed, n" signifies participants who were evaluable for this outcome measure at given time points.
Measure: Mean (Standard Deviation); unit: nanograms per milliliter (ng/mL)
Arm/Group | Treatment Arm A: Lenvatinib + Ifosfamide + Etoposide
Number analyzed (Participants) | 37
nanograms per milliliter (ng/mL)
  Cycle 1, Day 1: 0.5-4 hours post-dose | 147.9 (194.61)
  Cycle 1, Day 1: 6-10 hours post-dose: number analyzed (Participants) | 35
  Cycle 1, Day 1: 6-10 hours post-dose | 217.8 (99.54)
  Cycle 1, Day 15: Pre-dose: number analyzed (Participants) | 36
  Cycle 1, Day 15: Pre-dose | 70.7 (43.48)
  Cycle 1, Day 15: 0.5-4 hours post-dose | 222.3 (203.07)
  Cycle 1, Day 15: 6-10 hours post-dose: number analyzed (Participants) | 35
  Cycle 1, Day 15: 6-10 hours post-dose | 310.9 (106.79)
  Cycle 2, Day 1: Pre-dose | 70.2 (67.95)

10. Secondary Outcome: Change From Baseline in Pediatric Quality of Life Inventory (PedsQL) Scale: Generic Core Scale Score at Month 4
Description: Health-Related Quality of Life (HRQoL): PedsQL 4.0 Generic Core Scale is a multidimensional scale. It included assessment of 4 dimensions: physical functioning (8 items), emotional functioning (8 items), social functioning (8 items), and school functioning (5 items - children greater than or equal to [>=] 5 years, adults; 3 items - toddlers [aged 2-4 years]). Each item was reported using a 5-point Likert scale, items were then reverse-scored and linearly transformed to a 0 to 100 scale. Generic Core Scale total score: sum of all the items divided by the number of items answered across all the scales. Total score ranges from 0 to 100, where higher scores=better HRQoL, lower scores=worse HRQoL.
Time Frame: Baseline and Month 4
Population: HRQoL Analysis Set included all participants who had received at least 1 dose of study drug and had completed at least 1 postbaseline patient-reported outcome (PRO) assessment. Here "overall number of participants analyzed, N" signifies participants who were evaluable for this outcome measure.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Treatment Arm A: Lenvatinib + Ifosfamide + Etoposide | Treatment Arm B: Ifosfamide + Etoposide
Number analyzed (Participants) | 15 | 4
score on a scale | 2.61 (17.568) | 2.65 (4.128)

11. Secondary Outcome: Change From Baseline in PedsQL Scale: Cancer Module Scale Score at Month 4
Description: HRQoL: PedsQL 3.0 Cancer Module Scale measured pediatric cancer-specific HRQoL. It included assessment of 8 dimensions: pain and hurt (2 items), nausea (5 items), procedural anxiety (3 items), treatment anxiety (3 items), worry (3 items), cognitive problems (3 items - toddlers [aged 2-4], 4 items - young children [aged 5-7]; 5 items for children aged >=8 years, adults), perceived physical appearance (3 items), communication (3 items). Each item was reported using a 5-point Likert scale, items were then reverse-scored and linearly transformed to a 0 to 100 scale. Cancer Module total score: sum of all items divided by the number of items answered on all the scales. Total score ranges from 0 to 100, where higher scores=better HRQoL, lower scores=worse HRQoL.
Time Frame: Baseline and Month 4
Population: HRQoL Analysis Set included all participants who had received at least 1 dose of study drug and had completed at least 1 postbaseline PRO assessment. Here "overall number of participants analyzed, N" signifies participants who were evaluable for this outcome measure.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Treatment Arm A: Lenvatinib + Ifosfamide + Etoposide | Treatment Arm B: Ifosfamide + Etoposide
Number analyzed (Participants) | 16 | 4
score on a scale | 2.66 (9.989) | 2.08 (6.736)

12. Secondary Outcome: Number of Participants Categorized Based on Overall Palatability and Acceptability Questionnaire Responses for Suspension of Lenvatinib
Description: The palatability and acceptability of lenvatinib oral suspension formulation was assessed using the Palatability Questionnaire. In the questionnaire, participants were asked to answer palatability and acceptability of lenvatinib suspension considering the following elements: taste, appearance, smell, how does it feel in the mouth and overall acceptability in terms of 7 responses: Super good, really good, good, may be good or may be bad, bad, really bad, super bad. In this outcome measure, number of participants have been reported per their overall palatability and acceptability responses.
Time Frame: Cycle 1 Day 1 (Cycle length = 21 days)
Population: Palatability and acceptability analysis set included all participants who received oral suspension of lenvatinib in Treatment Arm A and who received an optional lenvatinib suspension in Treatment Arm B and who answered at least 1 question in the palatability questionnaire. As planned, combined data for Lenvatinib from Treatment Arm A and B was reported for this outcome measure. Here "overall number of participants analyzed, N" signifies participants who were evaluable for this outcome measure.
Measure: Count of Participants; unit: Participants
Groups:
- All Participants: Lenvatinib 14 mg/m^2: Participants received lenvatinib 14 mg/m^2 suspension, orally, once daily in continuous 21-day cycles until PD, development of unacceptable toxicity, participant request, withdrawal of consent, or discontinuation of study by the sponsor. Participants who were unable to swallow capsules received lenvatinib as an extemporaneous suspension prepared from the capsule.
Arm/Group | All Participants: Lenvatinib 14 mg/m^2
Number analyzed (Participants) | 5
Participants
  Super Bad | 0
  Really Bad | 0
  Bad | 0
  May be Good or May be Bad | 2
  Good | 2
  Really Good | 0
  Super Good | 1

ADVERSE EVENTS:
Time Frame: From first dose up to 30 days after the last dose of study drug (up to 40.8 months)
Description: Treatment Arm B safety data for Ifosfamide + Etoposide to Lenvatinib (optional) were reported separately. All randomized participants were monitored for death (all-cause mortality). Only treated participants were assessed for adverse events (serious and non-serious).
Groups:
- Treatment Arm B: Ifosfamide+Etoposide to Lenvatinib (Optional): Eligible participants from Treatment Arm B: Ifosfamide+Etoposide who had PD per RECIST v1.1 received an optional lenvatinib treatment (14 mg/m^2, capsules, orally, once daily in continuous 21-day cycles until next PD, development of unacceptable toxicity, participant choice, withdrawal of consent or discontinuation of study by the sponsor, whichever occurred first) plus any remaining cycles of chemotherapy if 5 cycles were not completed prior to PD.
Arm/Group | Treatment Arm A: Lenvatinib + Ifosfamide + Etoposide | Treatment Arm B: Ifosfamide + Etoposide | Treatment Arm B: Ifosfamide+Etoposide to Lenvatinib (Optional)
All-Cause Mortality (participants affected / at risk) | 25/40 | 25/41 | 12/16
Serious Adverse Events (participants affected / at risk) | 30/39 | 20/39 | 10/16
Other Adverse Events (participants affected / at risk) | 38/39 | 39/39 | 16/16
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment Arm A: Lenvatinib + Ifosfamide + Etoposide (N=39) | Treatment Arm B: Ifosfamide + Etoposide (N=39) | Treatment Arm B: Ifosfamide+Etoposide to Lenvatinib (Optional) (N=16)
Anaemia (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0)
Febrile neutropenia (Blood and lymphatic system disorders) | 15 (27) | 7 (10) | 0 (0)
Neutropenia (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0)
Thrombocytopenia (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0)
Cardiac failure (Cardiac disorders) | 1 (2) | 0 (0) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 2 (2) | 0 (0) | 0 (0)
Anal fistula (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 1 (1) | 0 (0) | 1 (1)
Nausea (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Stomatitis (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Vomiting (Gastrointestinal disorders) | 0 (0) | 1 (2) | 1 (1)
Catheter site ulcer (General disorders) | 1 (1) | 0 (0) | 0 (0)
Pyrexia (General disorders) | 6 (7) | 2 (3) | 1 (1)
Cholecystitis (Hepatobiliary disorders) | 1 (1) | 0 (0) | 0 (0)
Gallbladder obstruction (Hepatobiliary disorders) | 1 (1) | 0 (0) | 0 (0)
Hepatitis acute (Hepatobiliary disorders) | 1 (1) | 0 (0) | 0 (0)
Anaphylactic reaction (Immune system disorders) | 0 (0) | 1 (1) | 0 (0)
Drug hypersensitivity (Immune system disorders) | 0 (0) | 1 (1) | 0 (0)
Bacteraemia (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
COVID-19 (Infections and infestations) | 2 (3) | 0 (0) | 0 (0)
Device related infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Escherichia sepsis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Gastroenteritis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Infection (Infections and infestations) | 0 (0) | 1 (2) | 0 (0)
Infectious pleural effusion (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Osteomyelitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Pleural infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Pneumonia (Infections and infestations) | 2 (3) | 0 (0) | 1 (2)
Pneumonia fungal (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Post procedural cellulitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Respiratory syncytial virus infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Sepsis (Infections and infestations) | 0 (0) | 2 (3) | 0 (0)
Skin infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Staphylococcal sepsis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Vascular device infection (Infections and infestations) | 0 (0) | 2 (2) | 0 (0)
Wound infection staphylococcal (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Post procedural haemorrhage (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Postoperative wound complication (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Wound dehiscence (Injury, poisoning and procedural complications) | 2 (2) | 1 (1) | 0 (0)
Haemoglobin decreased (Investigations) | 0 (0) | 1 (2) | 0 (0)
Neutrophil count decreased (Investigations) | 1 (1) | 1 (1) | 0 (0)
Platelet count decreased (Investigations) | 3 (3) | 0 (0) | 0 (0)
Transaminases increased (Investigations) | 1 (1) | 0 (0) | 0 (0)
Decreased appetite (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0)
Dehydration (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0)
Hypokalaemia (Metabolism and nutrition disorders) | 1 (5) | 0 (0) | 0 (0)
Hypophosphataemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0)
Bone pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Cancer pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0)
Malignant pleural effusion (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 4 (6) | 1 (1) | 0 (0)
Metastases to central nervous system (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
Metastases to heart (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
Tumour pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0)
Malignant spinal cord compression (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Metabolic encephalopathy (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Posterior reversible encephalopathy syndrome (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Seizure (Nervous system disorders) | 2 (2) | 1 (1) | 0 (0)
Syncope (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Toxic encephalopathy (Nervous system disorders) | 3 (4) | 0 (0) | 0 (0)
Device breakage (Product Issues) | 0 (0) | 2 (2) | 0 (0)
Device extrusion (Product Issues) | 1 (1) | 0 (0) | 0 (0)
Cystitis haemorrhagic (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0)
Haematuria (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0)
Proteinuria (Renal and urinary disorders) | 2 (3) | 0 (0) | 0 (0)
Renal tubular injury (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 (2) | 1 (1) | 0 (0)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (2) | 0 (0)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 (2) | 1 (1) | 0 (0)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 7 (12) | 1 (1) | 4 (8)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1) | 0 (0)
Deep vein thrombosis (Vascular disorders) | 1 (1) | 1 (1) | 0 (0)
Hypertension (Vascular disorders) | 1 (1) | 0 (0) | 1 (1)
Hypertensive urgency (Vascular disorders) | 1 (1) | 0 (0) | 0 (0)
Constipation (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Pain (General disorders) | 0 (0) | 0 (0) | 1 (1)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Spinal cord compression (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Acute kidney injury (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (2)
Oedema peripheral (General disorders) | 0 (0) | 0 (0) | 1 (1)
Cholecystitis acute (Hepatobiliary disorders) | 0 (0) | 0 (0) | 1 (1)
Lower respiratory tract infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Pulmonary haemorrhage (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment Arm A: Lenvatinib + Ifosfamide + Etoposide (N=39) | Treatment Arm B: Ifosfamide + Etoposide (N=39) | Treatment Arm B: Ifosfamide+Etoposide to Lenvatinib (Optional) (N=16)
Anaemia (Blood and lymphatic system disorders) | 28 (180) | 27 (102) | 2 (10)
Febrile neutropenia (Blood and lymphatic system disorders) | 1 (1) | 4 (4) | 0 (0)
Leukopenia (Blood and lymphatic system disorders) | 5 (53) | 4 (27) | 2 (2)
Lymphopenia (Blood and lymphatic system disorders) | 1 (17) | 4 (26) | 0 (0)
Neutropenia (Blood and lymphatic system disorders) | 9 (39) | 9 (20) | 3 (3)
Thrombocytopenia (Blood and lymphatic system disorders) | 6 (50) | 5 (12) | 0 (0)
Tachycardia (Cardiac disorders) | 2 (3) | 3 (3) | 0 (0)
Hypothyroidism (Endocrine disorders) | 35 (52) | 0 (0) | 8 (9)
Hyperthyroidism (Endocrine disorders) | 3 (3) | 0 (0) | 0 (0)
Eye pain (Eye disorders) | 2 (4) | 0 (0) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 7 (18) | 3 (4) | 3 (12)
Abdominal pain upper (Gastrointestinal disorders) | 4 (6) | 1 (1) | 2 (3)
Constipation (Gastrointestinal disorders) | 14 (20) | 5 (6) | 4 (6)
Diarrhoea (Gastrointestinal disorders) | 14 (20) | 2 (2) | 4 (8)
Gastritis (Gastrointestinal disorders) | 0 (0) | 2 (2) | 0 (0)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 2 (2) | 0 (0) | 1 (1)
Mouth ulceration (Gastrointestinal disorders) | 1 (1) | 2 (2) | 1 (1)
Nausea (Gastrointestinal disorders) | 23 (56) | 16 (30) | 5 (6)
Proctalgia (Gastrointestinal disorders) | 3 (6) | 1 (1) | 0 (0)
Stomatitis (Gastrointestinal disorders) | 10 (14) | 6 (7) | 1 (3)
Toothache (Gastrointestinal disorders) | 2 (2) | 2 (2) | 0 (0)
Vomiting (Gastrointestinal disorders) | 19 (44) | 11 (17) | 5 (12)
Asthenia (General disorders) | 2 (2) | 0 (0) | 1 (1)
Face oedema (General disorders) | 2 (4) | 0 (0) | 0 (0)
Fatigue (General disorders) | 13 (28) | 9 (11) | 4 (8)
Generalised oedema (General disorders) | 1 (2) | 2 (3) | 0 (0)
Impaired healing (General disorders) | 2 (3) | 0 (0) | 0 (0)
Non-cardiac chest pain (General disorders) | 2 (3) | 0 (0) | 1 (1)
Oedema (General disorders) | 2 (2) | 0 (0) | 0 (0)
Pyrexia (General disorders) | 12 (16) | 5 (6) | 2 (2)
Hyperbilirubinaemia (Hepatobiliary disorders) | 3 (5) | 0 (0) | 0 (0)
COVID-19 (Infections and infestations) | 8 (9) | 1 (1) | 0 (0)
Catheter site infection (Infections and infestations) | 2 (2) | 0 (0) | 0 (0)
Hand-foot-and-mouth disease (Infections and infestations) | 2 (2) | 0 (0) | 0 (0)
Herpes zoster (Infections and infestations) | 2 (2) | 0 (0) | 0 (0)
Rash pustular (Infections and infestations) | 2 (2) | 0 (0) | 0 (0)
Rhinitis (Infections and infestations) | 4 (4) | 0 (0) | 0 (0)
Wound infection (Infections and infestations) | 2 (2) | 0 (0) | 0 (0)
Allergic transfusion reaction (Injury, poisoning and procedural complications) | 2 (2) | 0 (0) | 0 (0)
Procedural pain (Injury, poisoning and procedural complications) | 3 (6) | 0 (0) | 1 (1)
Alanine aminotransferase increased (Investigations) | 7 (27) | 4 (11) | 1 (1)
Amylase increased (Investigations) | 2 (2) | 0 (0) | 0 (0)
Aspartate aminotransferase increased (Investigations) | 7 (25) | 5 (11) | 3 (4)
Blood alkaline phosphatase increased (Investigations) | 3 (6) | 4 (5) | 1 (1)
Blood bicarbonate decreased (Investigations) | 0 (0) | 3 (7) | 0 (0)
Blood bilirubin increased (Investigations) | 3 (20) | 0 (0) | 0 (0)
Blood creatinine increased (Investigations) | 6 (9) | 0 (0) | 0 (0)
Blood lactate dehydrogenase increased (Investigations) | 1 (1) | 4 (4) | 1 (2)
Blood thyroid stimulating hormone increased (Investigations) | 5 (6) | 0 (0) | 3 (3)
C-reactive protein increased (Investigations) | 4 (4) | 0 (0) | 0 (0)
Ejection fraction decreased (Investigations) | 4 (5) | 0 (0) | 1 (1)
Electrocardiogram T wave abnormal (Investigations) | 2 (2) | 0 (0) | 0 (0)
Gamma-glutamyltransferase increased (Investigations) | 4 (18) | 2 (11) | 2 (2)
Lymphocyte count decreased (Investigations) | 5 (28) | 7 (32) | 1 (4)
Neutrophil count decreased (Investigations) | 15 (79) | 13 (38) | 1 (1)
Platelet count decreased (Investigations) | 23 (209) | 17 (57) | 3 (12)
SARS-CoV-2 test positive (Investigations) | 0 (0) | 2 (2) | 0 (0)
Weight decreased (Investigations) | 8 (13) | 4 (4) | 5 (10)
Weight increased (Investigations) | 2 (5) | 0 (0) | 0 (0)
White blood cell count decreased (Investigations) | 5 (38) | 13 (47) | 2 (8)
Decreased appetite (Metabolism and nutrition disorders) | 8 (10) | 5 (6) | 5 (10)
Dehydration (Metabolism and nutrition disorders) | 2 (3) | 1 (1) | 0 (0)
Hypervolaemia (Metabolism and nutrition disorders) | 2 (4) | 0 (0) | 0 (0)
Hypoalbuminaemia (Metabolism and nutrition disorders) | 4 (6) | 2 (2) | 1 (1)
Hypocalcaemia (Metabolism and nutrition disorders) | 2 (8) | 4 (9) | 1 (1)
Hypokalaemia (Metabolism and nutrition disorders) | 5 (19) | 6 (13) | 1 (1)
Hypomagnesaemia (Metabolism and nutrition disorders) | 6 (17) | 3 (5) | 2 (2)
Hyponatraemia (Metabolism and nutrition disorders) | 3 (4) | 3 (3) | 3 (3)
Hypophosphataemia (Metabolism and nutrition disorders) | 6 (26) | 7 (9) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 11 (24) | 6 (6) | 3 (4)
Back pain (Musculoskeletal and connective tissue disorders) | 15 (22) | 6 (7) | 4 (6)
Bone pain (Musculoskeletal and connective tissue disorders) | 4 (5) | 1 (1) | 1 (1)
Muscular weakness (Musculoskeletal and connective tissue disorders) | 2 (4) | 1 (1) | 1 (1)
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 5 (6) | 0 (0) | 0 (0)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 5 (6) | 1 (3) | 1 (1)
Myalgia (Musculoskeletal and connective tissue disorders) | 7 (15) | 0 (0) | 0 (0)
Neck pain (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 9 (14) | 5 (5) | 6 (21)
Trismus (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0) | 0 (0)
Malignant pleural effusion (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 (4) | 1 (1) | 0 (0)
Tumour pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (2) | 2 (3) | 0 (0)
Dizziness (Nervous system disorders) | 7 (8) | 2 (4) | 0 (0)
Headache (Nervous system disorders) | 14 (20) | 6 (6) | 5 (28)
Toxic encephalopathy (Nervous system disorders) | 2 (2) | 0 (0) | 0 (0)
Tremor (Nervous system disorders) | 3 (4) | 1 (1) | 0 (0)
Anxiety (Psychiatric disorders) | 3 (3) | 1 (1) | 1 (1)
Depression (Psychiatric disorders) | 3 (3) | 0 (0) | 1 (1)
Insomnia (Psychiatric disorders) | 3 (4) | 1 (1) | 2 (4)
Dysuria (Renal and urinary disorders) | 2 (2) | 1 (1) | 1 (1)
Glycosuria (Renal and urinary disorders) | 2 (2) | 4 (7) | 0 (0)
Haematuria (Renal and urinary disorders) | 4 (11) | 2 (2) | 0 (0)
Pollakiuria (Renal and urinary disorders) | 3 (3) | 0 (0) | 1 (1)
Proteinuria (Renal and urinary disorders) | 21 (79) | 5 (7) | 6 (21)
Cough (Respiratory, thoracic and mediastinal disorders) | 7 (7) | 5 (7) | 1 (2)
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0) | 1 (1)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 4 (6) | 3 (3) | 1 (1)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 12 (23) | 2 (2) | 0 (0)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 2 (3) | 0 (0) | 0 (0)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 4 (4) | 1 (1) | 1 (2)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0) | 0 (0)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 8 (19) | 1 (1) | 3 (7)
Alopecia (Skin and subcutaneous tissue disorders) | 3 (4) | 0 (0) | 0 (0)
Dry skin (Skin and subcutaneous tissue disorders) | 5 (6) | 1 (1) | 0 (0)
Palmar-plantar erythrodysaesthesia syndrome (Skin and subcutaneous tissue disorders) | 5 (11) | 0 (0) | 2 (2)
Rash (Skin and subcutaneous tissue disorders) | 8 (13) | 1 (1) | 1 (1)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 3 (3) | 1 (1) | 0 (0)
Urticaria (Skin and subcutaneous tissue disorders) | 5 (7) | 1 (1) | 0 (0)
Hypertension (Vascular disorders) | 16 (39) | 0 (0) | 6 (8)
Hypotension (Vascular disorders) | 2 (2) | 2 (2) | 0 (0)
Eosinophilia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1)
Pancytopenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1)
Angina pectoris (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
Cheilitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Dyspepsia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Gastrointestinal pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Early satiety (General disorders) | 0 (0) | 0 (0) | 1 (1)
Infusion site bruising (General disorders) | 0 (0) | 0 (0) | 1 (1)
Infusion site swelling (General disorders) | 0 (0) | 0 (0) | 1 (1)
Oedema peripheral (General disorders) | 0 (0) | 0 (0) | 1 (1)
Gingivitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Influenza (Infections and infestations) | 0 (0) | 0 (0) | 1 (2)
Muscle rupture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Blood magnesium decreased (Investigations) | 0 (0) | 0 (0) | 1 (1)
Blood pressure increased (Investigations) | 0 (0) | 0 (0) | 1 (2)
Haemoglobin increased (Investigations) | 0 (0) | 0 (0) | 1 (1)
Lipase increased (Investigations) | 0 (0) | 0 (0) | 2 (3)
Hypercalcaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 2 (3)
Cancer pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (2)
Aphasia (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Hypoaesthesia (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Lethargy (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Migraine (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Confusional state (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1)
Pharyngeal inflammation (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Pelvic pain (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 1 (1)
Hair colour changes (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Pain of skin (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Pruritus (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Rash macular (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Skin plaque (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Palpitations (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
Dry eye (Eye disorders) | 2 (2) | 1 (1) | 0 (0)
Aphthous ulcer (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Dry mouth (Gastrointestinal disorders) | 2 (2) | 0 (0) | 0 (0)
Cholecystitis acute (Hepatobiliary disorders) | 0 (0) | 0 (0) | 1 (1)
Overgrowth bacterial (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Paronychia (Infections and infestations) | 2 (3) | 1 (2) | 0 (0)
Vitamin D deficiency (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1)
Tumour haemorrhage (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (2)
Hypercholesterolaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1)
Hyperkalaemia (Metabolism and nutrition disorders) | 2 (2) | 1 (1) | 0 (0)
Duodenitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2020-09-10): https://cdn.clinicaltrials.gov/large-docs/89/NCT04154189/Prot_004.pdf
  • Statistical Analysis Plan (2022-06-15): https://cdn.clinicaltrials.gov/large-docs/89/NCT04154189/SAP_005.pdf